CLINICAL TRIAL: NCT01535378
Title: Interest of Behavioural Reeducation in Dysfunctions of Masticatory Apparatus. Relations Between Parafunctions and Dysfunctions of Mastixatory Apparatus
Acronym: PARADYSAM
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-A00838-33; LOC/11-06 (Other: Rennes University Hospital (Direction of Clinical Research))
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
If etiologies of temporomandibular disorders (TMD) are various, parafunctions become more and more important. Treatment of patients presenting TMD is based on conservative and reversible therapeutics. The behavioural reeducation of these patients which aims at decreasing their parafunctions is a treatment often performed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female over 18,
* Patient who was informed about the protocol and who did not refuse to take part in the programme,
* Patient who suffers of dysfunctions of masticatory apparatus: myofascial pain, joint clicking or crepitations, disc deplacement with reduction, mandibular limitation and/or deviation,
* Patient who presents more or less obvious parafunctions, which are associated or not to other etiologies
* Patient consulting for the 1st time for TMD

Exclusion Criteria:

* Persons over 18 who are under legal protection (guardianship), persons who are deprived of their freedom,
* Patient who is already followed in the consultation of dysfunctions of masticatory apparatus and who is under treatment,
* Patient who is under treatment of occlusal splint (not in the framework of the consultation of TMD
* Patient with pains other than orofacial pains (cephalalgia, neuralgia, vascular algia of the face, migraine),
* Patient who needs a treatment other than a behavioural reeducation (pharmacological treatment, occlusal splint , addressed to another therapist, prosthetic treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with temporomandibular disorders
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-03

PRIMARY OUTCOMES:
Assessment of pain based on the analogical visual scale | 1 year
  To know the incidence of a treatment which is unique, reversible and performed in first intention: behavioural reeducation in the evolution of clinical signs of TMD : pain; disc deplacement with reduction, limitation or mandibular deviation during mouth opening.

SECONDARY OUTCOMES:
Amplitude of mouth opening, mandibular deviation, joint clicking or crepitations,disc deplacement with reduction | 1 year
  Evaluation of parafunctions as an etiological factor of dysfunctions of masticatory apparatus.
Assessment of behavioural reeducation | 1 year
  Interest of diagnosis criteria of investigation on temporomandibular disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Chauvel-Lebret, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France